CLINICAL TRIAL: NCT01385956
Title: Phase I Study of Combination of SOM 230 Long Acting Release (LAR) + Gemcitabine in Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: SOM 230 and Gemcitabine in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16456; CSOM230CUS16T (Other: Norvartis)
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: metastatic; locally advanced; combination therapy; dose escalation; epithelial cancer; adenocarcinoma; exocrine pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — pasireotide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOM 230 LAR and Gemcitabine (Experimental): Combination Therapy: Dose escalation of SOM 230 LAR and standard treatment with gemcitabine. Treatment will be administered on an outpatient basis. Gemcitabine is administered by IV infusion. The dose should be based on the patient's actual baseline body weight; the dose will be recalculated if there is a weight change of > 10% from baseline. The dose of gemcitabine will be given over 30 minutes, weekly every 3 weeks followed by 1 week rest period.
  SOM 230 LAR will be administered as an intramuscular dose determined by the dosing schema, every month.
  Interventions: Drug: SOM 230 LAR; Drug: Gemcitabine

INTERVENTIONS:
Drug: SOM 230 LAR — We will attempt dose escalation starting at a lower level 1 of 40 mg since we are using SOM 230 LAR in combination with gemcitabine for the first time.
  Other Names: Pasireotide
Drug: Gemcitabine — Fixed dose: 1000mg/m^2 weekly x3 then 1 week off
  Other Names: Gemzar®)

SUMMARY:
The goal of this clinical research study is to learn if the study drug SOM 230 in addition to standard therapy of gemcitabine can shrink or slow the growth of pancreatic cancer. The safety and tolerability of different doses of SOM 230 will also be studied. The participants' physical state, changes in the size of the tumor, and laboratory findings taken while on-study will help us (the study doctor and Moffitt Cancer Center) decide if SOM 230 is safe and effective.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase I study of combination therapy with SOM 230 LAR and standard treatment with gemcitabine. We will utilize a staggered, sequential dose-escalation design to define the maximum tolerated dose (MTD) of SOM 230 LAR when combined with standard doses of gemcitabine. Cycle will be defined as 28 days.

Treatment will be administered on an outpatient basis. Gemcitabine is administered by IV infusion. The dose should be based on the patient's actual baseline body weight; the dose will be recalculated if there is a weight change of > 10% from baseline. The dose of gemcitabine will be given over 30 minutes, weekly every 3 weeks followed by 1 week rest period. SOM 230 LAR will be administered as an intramuscular dose determined by the dosing schema, every month.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed evidence of epithelial cancer (adenocarcinoma) of the exocrine pancreas
* Metastatic or locally advanced disease. Patients with measurable and with non measurable disease, as per RECIST criteria are eligible.
* Minimum of 4 weeks since any major surgery, completion of radiation
* Prior treatment with gemcitabine alone or 5-fluorouracil (5-FU) with radiation as an adjuvant therapy will be allowed if > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy ≥ 12 weeks
* Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L, Platelets ≥ 100 x 10^9/L, hemoglobin (Hgb) > 9 g/dL
* Adequate liver function as shown by: serum bilirubin ≤ 1.5 x upper limit of normal (ULN), and serum transaminases activity ≤ 3 x ULN, with the exception of serum transaminases (< 5 x ULN) if the patient has liver metastases.
* Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and WOCBP must be advised of the importance of using effective birth control measures during the course of the study.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.
* Screening electrocardiogram (ECG) with a time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole [QT] corrected for heart rate (QTc) < 450 msec

Exclusion Criteria:

* Prior treatment with any cytotoxic chemotherapy except as an adjuvant therapy
* Have undergone major surgery within 4 weeks prior to study enrollment
* Chronic treatment with steroids or any other immunosuppressant drugs
* Should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
* Untreated brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 1.5 ULN or glycosylated hemoglobin (HbA1c) >8%. Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted
* Patients with symptomatic cholelithiasis
* QT related exclusion criteria: Fridericia Correction Formula (QTcF) at screening > 450 msec; History of syncope or family history of idiopathic sudden death; Sustained or clinically significant cardiac arrhythmias; Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular (AV) block; Concomitant medication(s) known to prolong the QT interval (patient must be off the drug for 2 weeks to be eligible)
* Patients who have congestive heart failure [New York Heart Association (NYHA) Class III or IV], unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the 6 months preceding enrollment
* Known history of human immunodeficiency virus (HIV)
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Any active (acute or chronic) or uncontrolled infection/ disorders; Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (WOCBP must have a negative serum pregnancy test within 14 days prior to administration of pasireotide). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulations
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events | The end of each participant's 28 day cycle
  Safety / Tolerability (type, frequency, severity, and relationship of adverse events to study drug)

SECONDARY OUTCOMES:
Number of Participants With Progression Free Survival (PFS) | 3 months
  Frequency counts and percentage will be used to summarize the progression-free survival (PFS) in 3 months period.
Number of Participants With Tumor Response | 6 months
  Tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST). Objective tumor response will be summarized using frequency counts and percentage.
Number of Participants With Overall Survival (OS) | 6 months
  Frequency counts and percentage will be used to summarize the overall survival (OS) in 6 months period.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Suleiman Y, Mahipal A, Shibata D, Siegel EM, Jump H, Fulp WJ, Springett GM, Kim R. Phase I study of combination of pasireotide LAR + gemcitabine in locally advanced or metastatic pancreatic cancer. Cancer Chemother Pharmacol. 2015 Sep;76(3):481-7. doi: 10.1007/s00280-015-2814-8. Epub 2015 Jul 1. PMID 26126727